CLINICAL TRIAL: NCT03913858
Title: Does Low Flow Anesthesia Protect Lung Functions in Laparoscopic Sleeve Gastrectomy?
Brief Title: Low Flow Anesthesia in Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Evrim Kucur Tulubas, Department of Anesthesiology and Critical Care Medicine Attending Anaesthesia, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Obesity Surgery FEV1/FVC; Evrim Kucur Tulubas (Other: Bakirkoy Dr. Sadi Konuk Training and Research Hospital)
Record Dates: First submitted 2019-02-21; First posted 2019-04-12 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Morbid Obesity; Anesthesia Complication; Anesthesia; Functional
Keywords: Morbid Obesity; Sleeve Gastrectomy; Low Flow Anesthesia
MeSH Terms: conditions — Obesity, Morbid | interventions — Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-flow anesthesia (Other): Before beginning induction, first 3 mg midazolam and fentanyl 150 mvq IV were administered. According to ideal weight and BIS score for 40-60, 2-5 mg propofol and 0.5 mg rocuronium according to true weight were administered. After intubation 50 mg ranitidine and 8 mg ondansetron were routinely administered. Fixing the remifentanil dose to 0.1 mcg/kg/min, infusion was administered. Group 1 had 4 liter/minute (50% O2, 50% air) flow administered. Mechanical ventilator settings were 6-10 ml tidal volume, frequency 12/min (increasing, if necessary, for etCO2 35-45 mmHg), PEEP 5-10 cm/H2O and inspirium/expirium ratio ½. Both groups had remifentanil ended 10 minutes before the end of surgery. Later 1 g paracetamol and 100 mg tramadol IV were administered.
  Interventions: Procedure: Obesity Surgery with High-Flow Anesthesia
- low-flow anesthesia (Other): Before beginning induction, first 3 mg midazolam and fentanyl 150 mvq IV were administered. According to ideal weight and BIS score for 40-60, 2-5 mg propofol and 0.5 mg rocuronium according to true weight were administered. After intubation 50 mg ranitidine and 8 mg ondansetron were routinely administered. Fixing the remifentanil dose to 0.1 mcg/kg/min, infusion was administered. Group 2 had 1 liter/minute (50% O2, 50% air) flow administered. Mechanical ventilator settings were 6-10 ml tidal volume, frequency 12/min (increasing, if necessary, for etCO2 35-45 mmHg), PEEP 5-10 cm/H2O and inspirium/expirium ratio ½. Both groups had remifentanil ended 10 minutes before the end of surgery. Later 1 g paracetamol and 100 mg tramadol IV were administered.
  Interventions: Procedure: Obesity Surgery with Low-Flow Anesthesia

INTERVENTIONS:
Procedure: Obesity Surgery with Low-Flow Anesthesia — Group 1 had 1 liter/minute (50% O2, 50% air) flow administered.
  Other Names: Procedure/Anesthesia
  Arms: low-flow anesthesia
Procedure: Obesity Surgery with High-Flow Anesthesia — Group 2 had 4 liter/minute (50% O2, 50% air) flow administered.
  Other Names: Procedure/Anesthesia
  Arms: high-flow anesthesia

SUMMARY:
In this study to planned to research the efficacy of low-flow anesthesia on patients undergoing sleeve gastrectomy due to morbid obesity on respiratory functions after surgery by examining FEV1 and FVC values and FEV1/FVC ratio.

DETAILED DESCRIPTION:
Morbid obese patients undergoing sleeve gastrectomy due to morbid obesity after 01.01.2019 will be randomly divided into 2 groups with controls. To prevent selection bias in the study, numbers will be produced at random. The produced numbers will be determined as 0: control and 1: experiment groups and patients will be divided into groups as such. Random numbers will be generated by the MedCalc 18.2.1. program (MedCalc Statistical Software MedCalc Software bvba, Ostend, Belgium; http://www.medcalc.org; 2018). Group 1 is determined as patients to be administered high-flow anesthesia, while Group 2 will be administered low-flow anesthesia. After anesthesia induction, Group 1 will have 4 liters/minute (50% O2 50%) flow administered, while patients in Group 2 will have 1 liter/minute (50% O2, 50% air) flow administered. The study included adult patients who signed the voluntary consent form aged from 18-65 years, American Society of Anesthesiologists (ASA) III, and body mass index (BMI) >40. Inclusion criteria for the study are no alcohol or drug addiction or diagnosis of chronic obstructive pulmonary disease (COPD) during routine preoperative assessment by chest diseases, FEV1/FVC ratio, FEV1 and FVC values within normal limits and no previous abdominal surgery.

Those with stop-bang score below 4 will be included in the study. On the day of surgery, all patients had FEV1, FVC value and FEV1/FVC ratio examined by a single anesthesia technician using a manual RST device without the knowledge of the anesthesia expert.

Pressure tests and calibration of the anesthesia device is performed each morning for every surgery. After calibration the mechanical ventilator alarm limits for ins O2 are lower limit 40%, EtCO2 35-45 mmHg, min Vol (tidal volume in 1 min x frequency) according to the patient ± 0.5. After patient is placed on the operating table in ramp position, all patients are monitored with triple route ECG, pulse oximetry and pressure cuff. The clinical protocol for all patients undergoing sleeve gastrectomy includes BIS (bispectral index) and TOF (train of four) monitoring. Before beginning induction, first 3 mg midazolam and fentanyl 150 mvq IV were administered. According to ideal weight and BIS score for 40-60, 2-5 mg propofol and 0.5 mg rocuronium according to true weight were administered. Patients were ventilated with 6 L/min 60% O2 for 2 minutes. Patients were endotracheally intubated with a Macintosh laryngoscope. In addition to assessment of respiratory sounds linked to obesity with auscultation, EtCO2 capnography was used to confirm the efficacy of intubation. After intubation 50 mg ranitidine and 8 mg ondansetron were routinely administered. Fixing the remifentanil dose to 0.1 mcg/kg/min, infusion was administered. Sevoflurane percentage was changed to ensure MAC (minimum alveolar concentration of 0.6-1.1 for BIS score of 40-60 for maintenance. During ventilation in PRVC mode, Group 1 had 4 liter/minute (50% O2, 50% air) flow administered, while Group 2 had 3 L/min 4% for Sevoflurane the first 3 minutes as wash-in. Then flow was administered at 1 L/min (50% O2, 50% air). According to ideal weight, mechanical ventilator settings were 6-10 ml tidal volume, frequency 12/min (increasing, if necessary, for etCO2 35-45 mmHg), PEEP 5-10 cm/H2O and inspirium/expirium ratio ½. In Group 1, sevoflurane percentage was set to correlate with BIS monitoring. In Group 2, after intubation the sevoflurane percentage was set to a higher percentage to reach the desired MAC value. Every 5 minutes during surgery, MAC, BIS, mean arterial pressure, peak heart rate, sPO2, etCO2, inSO2, frequency and PEEP values were recorded. In Group 2, 5 minutes before the end of surgery, flow was increased from 1 L to 4 L for wash-out. Both groups had remifentanil ended 10 minutes before the end of surgery. Later 1 g paracetamol and 100 mg tramadol IV were administered. Five minutes before the end of the operation patient-controlled SIMV+VE mode with trigger setting of 6 was organized. At the end of surgery, patients were administered 2 mg/kg sugammadex according to ideal weight. When the patients trigger setting reaches muscle power it was lowered to zero. When trigger is zero and there is sufficient tidal volume to reach TOF (train of four) value >90% and BIS score is 80-100, patients were extubated. They were sent to the recovery room. In recovery the ARISCAT risk index was calculated. Later when modified Aldrete scoring system is ≥9, patients were sent to the ward.

After surgery, mobilization and respiratory physiotherapy were provided in the 2nd hour. Vital signs including mean arterial pressure (MAP) were recorded in the postoperative period with 20 mg tenoxicam I.V. administered in the 1st hour. The PCA device was set with tramadol 300 mg/100 ml, bolus 10 mg, lock time 12 minutes without basal infusion. Patients with numeric rating scale (NRS) scores ≥4 had a rescue dose of 4 mg morphine I.V. administered. Each patient began oral intake (water) in the postoperative 24th hour, with early mobilization. A second dose of tenoxicam I.V. was administered in the postoperative 8th hour.

In the 24th hour postoperative, patients had analgesia to ensure VAS score is below 4, with RFT repeated by the same doctor who performed RFT preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* american Society of Anesthesiologists (ASA) III
* body mass index (BMI) >40.
* FEV1/FVC ratio within normal limits
* FEV1 and FVC values within normal limits
* those with stop-bang score below 4

Exclusion criteria:

* alcohol abuse
* drug abuse
* previous abdominal surgery.
* chronic obstructive pulmonary disease (COPD)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Test Results | Preoperative 1st hour and postoperative 24th hours
  FEV1/FVC (%) ratio in hundred morbid obese patients who will undergo laparoscopic sleeve gastrectomy under low flow and high flow anesthesia will be measured

SECONDARY OUTCOMES:
Length of hospital stay | Up to 72th hours
  Length of hospital stay (days) of hundred morbid obese patients who will undergo laparoscopic sleeve gastrectomy under low flow and high flow anesthesia will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Kucur Tulubas, Dr, Principal Investigator
Locations (1):
- Bakırköy Dr. Sadi Konuk Trainig And Research Hospital, Istanbul, Turkey (Türkiye)